CLINICAL TRIAL: NCT00172705
Title: Quantitative Diagnosis of Fatty Liver by Dual Energy CT Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701262
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-02

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This study is proposed to explore the correlation between fatty content of fatty liver and the difference of CT attenuation value in men using dual-energy CT, and to set up a threshold for diagnosis of fatty liver.

DETAILED DESCRIPTION:
This study is proposed to explore the correlation between fatty content of fatty liver and the difference of CT attenuation value in men using dual-energy CT, and to set up a threshold for diagnosis of fatty liver.

ELIGIBILITY:
Inclusion Criteria:

* hepatic tumor
* living liver donor

Exclusion Criteria:

* pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-09; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: HON-MAN LIU, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Province of Taiwan, Taiwan